CLINICAL TRIAL: NCT07075380
Title: National Survey on Physical and Sports Activity of Adults With Epilepsy
Acronym: ENAPSE
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: NMR_2025_3
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with epilepsy
  Interventions: Behavioral: online questionnaire

INTERVENTIONS:
Behavioral: online questionnaire — Online questionnaire assessing physical activity level, completed twice at a 6-month interval.

SUMMARY:
Epilepsy affects nearly 600,000 people in France and causes neurological seizures that can lead to lasting impairments and stigma. Physical activity provides many benefits, including improved quality of life, social participation, and reduced stress and seizure frequency. Despite these benefits, people with epilepsy tend to be less active than the general population due to barriers such as fear of seizures during exercise, fatigue, and negative beliefs about the disease. Psychological factors and stigma influence physical activity engagement and affect how the disease is integrated into personal identity, impacting quality of life and treatment adherence. Studying the role of anxiety, stigma, and illness identity, as well as their interaction with physical activity identity, is essential to better understand and promote physical activity among people with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals self-reporting as over 18 years old
* Individuals self-reporting having epilepsy

Exclusion Criteria:

* not having completed secondary questionnaire at 6 months from inclusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Epileptic person willing to complete an online questionnaire about their physical activity
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
maintained physical activity | Day 0 and Month 6
  Physical activity level will be measured using an adapted version of the Modifiable Activity Questionnaire (MAQ) at inclusion and 6 months later as a criterion for behavior maintenance. MAQ ranges starts from 0 with no maximum limit. A higher value means a higher physical activity level.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut La Teppe, Tain-l'Hermitage, France